CLINICAL TRIAL: NCT05123157
Title: Pattern and Type of Amputation and Mortality Rate Associated With Diabetic Foot in Jeddah, Saudi Arabia: A Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Abdullah Abdulaziz Almohammadi, Doctor, King Abdulaziz University
Other Study IDs: 465- 20
Record Dates: First submitted 2021-10-20; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Foot; Amputation
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NO intervention — N/:
  NO intervention

SUMMARY:
This study explored the pattern and type of amputations performed on patients with diabetic foot who were admitted to our institution, as well as the 7-year mortality rate of patients with diabetic foot at the same institution. We believe that our study makes a significant contribution to the literature because it highlights the need for strengthening efforts to decrease the risk of amputation and mortality among patients with diabetic foot, especially in Jeddah, Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

* From the medical records of King Abdulaziz University Hospital (KAUH).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: medical records of King Abdulaziz University Hospital (KAUH).
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Rate and Pattern of amputation. | 7 years
  identify how many patients with Diabetic foot underwent amputation, and what type of amputation (major or minor)
Mortality among patients with diabetic foot | 7 years
  7-years mortality rate and predictive variable of death among patients with Diabetic foot.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No